CLINICAL TRIAL: NCT03023397
Title: Evaluation of the Effect of a Nasal Allergen Challenge With Dermatophagoides Farinae Extract on Nasal Airway Inflammation in Allergic Individuals, Comparing E-cigarette Users to Cigarette Smokers and Non-smokers.
Acronym: Mitey Nose
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1622; P50HL120100-05 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Healthy Participants; Tobacco Smokers
Keywords: E-cig smokers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Der f treated Non-smoker (Other)
  Interventions: Biological: Der f
- Der f treated Cigarette smoker (Other)
  Interventions: Biological: Der f
- Der f treated E-cig user (Other)
  Interventions: Biological: Der f

INTERVENTIONS:
Biological: Der f — Nasal administration of Dermatophagoides farinae with 100 allergen units (AU), 500 AU, and finally 1000 AU
  Other Names: (Der f)

SUMMARY:
The purpose of this pilot study is to evaluate allergen-induced nasal airway inflammation following nasal application of Dermatophagoides farinae (Der f), or house dust mite, extract in e-cigarette users, cigarette smokers, and non-smokers.

DETAILED DESCRIPTION:
The recent increase in popularity of e-cigarettes for smoking cessation or in combination with conventional cigarettes has led to safety concerns regarding their potential role in respiratory disease. These tobacco alternative devices were initially perceived as a "safer" alternative to cigarettes and were marketed without much known about their health effects. Increasing evidence demonstrates that while they contain fewer toxins and carcinogens than conventional cigarettes, they do involve delivery of ultrafine particles to the lower airways and can contain heavy metals and other chemicals. Tobacco smoke may augment allergic inflammation resulting from allergic rhinitis and/or asthma. Animal models of allergic asthma demonstrate aggravation of allergen-induced airway inflammation following inhalation of e-cig cartridge solution, with increased airway eosinophil infiltration, production of Th2 cytokines, and airway hyperresponsivness. In vitro studies in human tissues have demonstrated pro-inflammatory responses to e-cig vapour extract yet have not evaluated the effects of e-cig usage on allergic inflammation in human airways. Current evidence suggests that e-cigarette use augments allergic inflammatory responses in a similar way as tobacco smoke, yet a head-to-head comparison of the effects of these two exposures has not been performed in humans.

Use of tobacco products remains a pervasive problem in our society and around the world, with significant impact on respiratory health and quality of life. With the emergence of new non-tobacco based nicotine products like e-cigarettes, it is important to understand the impact these substances have on respiratory health and disease. The aim of this study is to study the impact of these products on allergic inflammation in house dust mite-allergic subjects who already routinely use e-cigarettes and to compare their responses to those of cigarette smokers and non-smokers. A thorough understanding of the potential health impacts of tobacco alternative substances is needed, especially given the rising popularity of such products with adolescents and young adults to whom these substances have particular appeal given their purported "safety" and variety of flavors to choose from.

ELIGIBILITY:
Inclusion Criteria:

1. Specific allergy to house dust mite D. farinae confirmed by positive immediate skin test response
2. Subjects will either be non-asthmatic or have mild asthma characterized by an Forced expiratory volume in one second (FEV1) of at least 80% of predicted to Forced vital capacity (FVC) ratio of at least .75
3. Subjects will be classified as tobacco smokers, e-cigarette users, or non-smokers according to the following guidelines.
4. Ability to withhold antihistamine medications for one week prior to baseline and allergen challenge visits
5. Subjects must be able and willing to give informed consent.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the allergen challenge study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, bleeding disorder, or chronic thyroid disease.
2. Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months.
3. Use of systemic steroid therapy within the preceding 12 months for treatment of an asthma exacerbation.
4. Use of inhaled or nasal steroids, cromolyn or leukotriene receptor antagonists (Montelukast or zafirlukast ) within the past month (except for use of cromolyn exclusively prior to exercise).
5. Subjects who smoke marijuana or use illicit drugs will be excluded.
6. Use of daily theophylline within the past month.
7. Use of nasal medications that might alter the response to nasal allergen challenge including anti-inflammatory and anti-histamine agents within one week of challenge.
8. Inability to withhold inhaled or oral bronchodilator medications for 12 hours prior to allergen challenge.
9. Pregnancy or nursing a baby.
10. Women of child-bearing age who are not using dependable contraception (such as birth control pills, intrauterine device (IUD), estrogen patches) or who are not completely abstinent.
11. Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
12. Exacerbation of asthma more than 2x/week which would be characteristic of a person with moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
13. Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
14. Viral upper respiratory tract infection or other acute inflammatory conditions of the nose or paranasal sinuses, such as sinusitis, within 4 weeks of challenge.
15. Any acute infection requiring antibiotics within 4 weeks of challenge.
16. Participating in an allergen inhalation study within 2 weeks of this challenge or use of any other investigational agent within the last 30 days.
17. Use of tricyclic antidepressants or beta-blockers.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from individuals who completed the general screening process at the Center for Environmental Medicine, Asthma and Lung Biology.
Groups:
- Non-smokers: Non-smoking adults with a history of dust mite allergy and allergic rhinitis
- Cigarette Smokers: Cigarette smoking adults with a history of dust mite allergy and allergic rhinitis
- E-cig Users: E-cig using adults with a history of dust mite allergy and allergic rhinitis
Period: Run-In
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Started | 8 | 3 | 1
Completed | 6 | 3 | 1
Not Completed | 2 | 0 | 0
Not completed — Failed screening allergen challenge | 1 | 0 | 0
Not completed — Loss of funding after informed consent but before screening allergen challenge | 1 | 0 | 0
Period: Main Study
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Started | 6 | 3 | 1
Completed | 6 | 3 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users | Total
Number analyzed (Participants) | 8 | 3 | 1 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 1 | 12
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 29.6 [20.1 to 35] | 34.6 [28.5 to 41.1] | 21.4 [21.4 to 21.4] | 29 [20.1 to 41.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 7
  Male | 3 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 7 | 2 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 0 | 5
  White | 5 | 1 | 1 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 3 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Eosinophils Per mL in Nasal Lavage Fluid (NLF)
Description: NLF will be collected immediately prior to administration of the nasal allergen challenge and 4 hours after completion of nasal allergen challenge. The protocol was amended to replace this outcome using Eosinophilic Cationic Protein (ECP) in Nasal Epithelial Lining Fluid (NELF).
Time Frame: Baseline, 4 hours post-allergen challenge
Population: NLF samples obtained from six non-smokers, 3 smokers and 1 e-cig user were contaminated with blood and therefore were not suitable samples for analysis of nasal inflammatory cells. The protocol was changed to include eosinophilic cationic protein (ECP) in nasal epithelial lining fluid (NELF) as the primary outcome measure.
Groups:
- Non-smokers: Intranasal administration of Dermatophagoides farinae allergen is performed until the participant reaches a total nasal symptom score (TNSS) of 8 or more AND a reduction in peak nasal inspiratory flow (PNIF) of 20% or more (or until the highest allergen dose is administered).
- Cigarette Smokers; E-cig Users: Intranasal administration of Dermatophagoides farinae allergen is performed until the participant reaches a TNSS of 8 or more AND a reduction in PNIF of 20% or more (or until the highest allergen dose is administered).
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Mean Change in Eosinophilic Cationic Protein (ECP) Levels in Nasal Epithelial Lining Fluid (NELF)
Description: NELF will be collected immediately prior to administration of the nasal allergen challenge and 4 hours after completion of nasal allergen challenge.
Time Frame: baseline, 4 hours post-allergen challenge
Population: Six non-smoking participants, 3 smoking participants and 1 e-cig using participant had paired pre and 4 hours post-challenge samples for analysis.
Measure: Mean (Standard Deviation); unit: micrograms/L
Groups:
- Non-smokers; Cigarette Smokers; E-cig Users: Intranasal administration of Dermatophagoides farinae allergen is performed until the participant reaches a TNSS of 8 or more AND a reduction in PNIF of 20% or more (or until the highest allergen dose is administered).
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 6 | 3 | 1
micrograms/L | 31374 (37261) | -50847 (45535) | -17851 (0)

3. Secondary Outcome: Mean Change in Interleukin-31 (IL-31) Concentrations in NELF
Description: NELF will be collected immediately prior to administration of the nasal allergen challenge, and 4 hours post- nasal allergen challenge.
Time Frame: Pre- and 4 hours-post nasal allergen challenge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 6 | 3 | 1
picograms/mL | 0.76 (1.01) | 0.06 (0.28) | 4.76 (0)

4. Secondary Outcome: Mean Change in Interleukin-5 (IL-5) Concentrations in NELF
Description: as for outcome 3
Time Frame: baseline, 4 hours post-allergen challenge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 6 | 3 | 1
picograms/mL | 75.82 (53.02) | 3.42 (4.58) | 240.9 (0)

5. Secondary Outcome: Mean Change in Macrophage Inflammatory Protein 1 Alpha (MIP-1a) Concentration in NELF
Description: as for outcome 3
Time Frame: baseline, 4 hours post-allergen challenge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 6 | 3 | 1
picograms/mL | 72.52 (42.9) | 10.04 (8.03) | 91.43 (0)

6. Secondary Outcome: Mean Change in Macrophage Inflammatory Protein 1 Beta (MIP-1b) in NELF
Description: as for outcome 3
Time Frame: baseline, 4 hours post-allergen challenge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 6 | 3 | 1
picograms/mL | 370.8 (511.6) | 18.97 (12.01) | 32.98 (0)

7. Other Pre Specified Outcome: Nasal Epithelial Cell Messenger Ribonucleic Acid (mRNA) Expression
Description: Nasal epithelial cell biopsies will be collected at baseline and 4 hours post- nasal allergen challenge. Gene expression changes will be quantified using quantitative real-time polymerase chain reaction (qRT-PCR).
Time Frame: Baseline, 4 hours post- nasal allergen challenge
Population: No samples were analyzed due to lack of funding and early termination of the study
Arm/Group | Non-smokers | Cigarette Smokers | E-cig Users
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of informed consent to the final study visit (up to 6 months).
Groups:
- Non-smoker: Non-smoking adults with a history of dust mite allergy and allergic rhinitis
- Cigarette Smoker: Cigarette smoking adults with a history of dust mite allergy and allergic rhinitis
- E-cig User: E-cig using adults with a history of dust mite allergy and allergic rhinitis
Arm/Group | Non-smoker | Cigarette Smoker | E-cig User
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 4/8 | 0/3 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-smoker (N=8) | Cigarette Smoker (N=3) | E-cig User (N=1)
Epistaxis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) — Mild epistaxis post nasal lavage administration - self resolved.
Headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Headache post nasal allergen challenge
Rhinitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) — Continued rhinitis experienced within 96 hours of nasal allergen challenge
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — non-productive cough 30 minutes post nasal allergen challenge administration
Sneeze (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Continued sneezing within 96 hours of nasal allergen challenge

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT03023397/Prot_SAP_000.pdf